CLINICAL TRIAL: NCT06533397
Title: The Application of a Biphasic Calcium Sulfate Graft Material in Sinus Floor Elevation
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Semmelweis University (Other)
Responsible Party: Principal Investigator, Marton Kivovics, associate professor, Semmelweis University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SEDCD44
Record Dates: First submitted 2024-07-24; First posted 2024-08-01 (Actual); Last update posted 2024-11-29 (Actual); Status verified 2024-08

CONDITIONS: Alveolar Bone Loss; Edentulism Nos
Keywords: bone graft material; biphasic calcium sulfate; sinus floor elevation; sinus lift; maxillary sinus augmentation; microcomputed tomography; cone beam computed tomography; histology; histomorphometry; dental implant
MeSH Terms: conditions — Alveolar Bone Loss | interventions — Sinus Floor Augmentation; formycin diphosphate; Bone Transplantation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- 3-month healing period (Experimental): Staged SFE is performed; following a 3-month-long healing period, bone core biopsy samples are harvested from the augmented bone, and dental implants are placed.
  Interventions: Procedure: Sinus floor elevation (SFE); Diagnostic Test: preoperative cone beam computed tomography (CBCT); Diagnostic Test: postoperative CBCT; Diagnostic Test: bone core biopsy; Procedure: dental implant placement; Procedure: fixed dental prosthesis (FDP) fabrication; Device: bone grafting
- 6-month healing period (Experimental): Staged SFE is performed; following a 6-month-long healing period, bone core biopsy samples are harvested from the augmented bone, and dental implants are placed.
  Interventions: Procedure: Sinus floor elevation (SFE); Diagnostic Test: preoperative cone beam computed tomography (CBCT); Diagnostic Test: postoperative CBCT; Diagnostic Test: bone core biopsy; Procedure: dental implant placement; Procedure: fixed dental prosthesis (FDP) fabrication; Device: bone grafting

INTERVENTIONS:
Procedure: Sinus floor elevation (SFE) — Patients rinse with 0.2% chlorhexidine solution for one minute before surgery. Under local anesthesia, a mucoperiosteal flap is raised from a midcrestal incision and two relieving incisions. Lateral window osteotomies are carried out using diamond burs. The Schneiderian membrane is carefully elevated and the synthetic bone graft material (Bond Apatite, Augma Biomaterials, Cesarea, Israel) (2-3 cm3) is packed in the defect with light force. The buccal flap is then mobilized to allow tension-free primary closure. The margins are stabilized with single interrupted sutures. Antibiotics (1 g amoxicillin-clavulanate twice a day for 5 days, or in case of side effects or known allergy to penicillin, 300 mg clindamycin 4 times a day for 4 days), anti-inflammatory drugs (50 mg diclofenac 3 times a day for 3 days), and chlorhexidine mouthwash (twice a day for 21 days from the first day after surgery) are prescribed. Suture removal takes place after 10 days.
  Other Names: sinus lift surgery; maxillary sinus augmentation
Diagnostic Test: preoperative cone beam computed tomography (CBCT) — A CBCT scan is performed before SFE surgery to evaluate the anatomy and pathologies of the maxillary sinus.
Diagnostic Test: postoperative CBCT — A CBCT scan is performed following the 3- or 6-month-long healing period after SFE to evaluate the anatomy and healing of the augmented bone and the maxillary sinus.
Diagnostic Test: bone core biopsy — At the time of dental implant placement, the first step of the implant bed preparation is performed using a trephine drill to harvest a bone core biopsy sample from the augmented bone. The biopsy sample is harvested from the implant bed, this way the patient is spared of excess surgical burden as this bone would be removed even if no biopsy sample was harvested during dental implant placement. The bone core biopsy samples are subjected to histomorphometric and microCT analysis.
Procedure: dental implant placement — Following the 3- or 6-month-long healing period following SFE, dental implants are placed non-submerged in the augmented bone under local anesthesia.
Procedure: fixed dental prosthesis (FDP) fabrication — 3 months after dental implant placement, fixed dental prostheses are delivered on the dental implants.
Device: bone grafting — A synthetic bone graft material (Bond Apatite, Augma Biomaterials, Cesarea, Israel) is used during SFE.

SUMMARY:
Pneumatization of the maxillary sinus may lead to insufficient bone volume for dental implant placement in the edentulous posterior maxilla. Sinus floor elevation (SFE) surgery with the lateral window technique is a safe and predictable surgical intervention to restore bone height in the maxillary premolar and molar areas. According to the literature, several bone graft materials may be successfully applied for SFE surgery. There is a lack of evidence regarding the application of biphasic calcium sulfate (BCS) for SFE. The healing period following staged SFE is 2-9 months.

The aim of this study is:

* to evaluate the success of SFE surgery using BCS as graft material,
* to compare the microarchitecture of the augmented bone depending on the healing period,
* to evaluate the success of dental implants placed in the augmented bone and that of the prostheses delivered on the dental implants.

ELIGIBILITY:
Inclusion Criteria:

* Patients over the age of 18 years,
* Patients who need dental implant-borne prostheses,
* Patients with insufficient bone height in the posterior maxilla due to sinus pneumatization.

Exclusion criteria:

.• Patients who had major systemic diseases as classified by the American Society of Anesthesiologists (ASA grades III-IV),

* psychiatric contraindications,
* patients on medication interfering with bone metabolism, including steroid therapy and antiresorptive medication,
* radiation to the head or neck region within the previous five years,
* localized periapical disease, odontogenic and nonodontogenic cysts, and maxillary sinusitis,
* evidence of uncontrolled periodontal disease,
* Alcohol Use Disorder defined by the Diagnostic and Statistical Manual of Mental Disorders, 5th Edition (DSM-5),
* recreational drug abuse,
* heavy smoking (>10 cigarettes/day),
* diseases of the oral mucosa, including blisters and ulcers, i.e.: red and white lesions, pigmented lesions, benign tumors of the oral cavity, and oral cancer. Leukoplakia, Erythroplakia, Precancerous lesions, Oral squamous cell carcinoma and malign tumors of the soft and hard tissues, Oral candidiasis, Oral lichen planus, Psoriasis, Pemphigus, and Pemphigoid.
* pregnancy or nursing,
* poor oral hygiene

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-08-24 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2031-09 (Estimated)

PRIMARY OUTCOMES:
Success of the SFE | 3 or 6 months
  The SFE surgery is successful if no inflammatory complications occur in the 3- or 6-month-long healing period and the bone volume is sufficient for dental implant placement.
Success of the dental implants | 5 years
  According to The International Congress of Oral Implantologists (ICOI) Pisa Consensus Conference.
  Success (optimum health)
  1. No pain or tenderness upon function
  2. 0 mobility
  3. less than 2 mm radiographic bone loss from initial surgery
  4. No exudates in the patient's history
  II. Satisfactory survival
  1. No pain on function
  2. 0 mobility
  3. 2-4 mm radiographic bone loss
  4. No exudates in the patient's history
  III. Compromised survival
  1. May have sensitivity on function
  2. No mobility
  3. Radiographic bone loss of more than 4 mm (less than1/2 of the length of the implant body)
  4. Probing depth more than 7 mm
  5. May have exudates in the patient's history
  IV. Failure (clinical or absolute failure)
  Any of the following:
  1. Pain on function
  2. Mobility
  3. Radiographic bone loss of more than 1/2 length of the implant
  4. Uncontrolled exudate
  5. Implant no longer in mouth
Success of the implant borne prostheses | 5 years
  Prostheses with four or fewer complications (screw loosening, decementation, chipping) that could be treated chairside.

SECONDARY OUTCOMES:
Hisomorphometry: Percent of residual bone graft particles | 3-6 months
  The percentage of residual bone graft particle-area measured on the representative sections prepared from the bone core biopsy samples. Unit: percent (%)
Hisomorphometry: Percent of newly formed bone | 3-6 months
  The percentage of newly formed bone-area measured on the representative sections prepared from the bone core biopsy samples. Unit: percent (%)
Hisomorphometry: Percent of bone marrow | 3-6 months
  The percentage of bone marrow-area measured on the representative sections prepared from the bone core biopsy samples. Unit: percent (%)
Value of the percent bone volume (BV/TV) calculated from the microCT reconstructions of the bone core biopsy samples. | 3-6 months
  Relative volume of calcified tissue in the selected volume. Unit: none
Value of the bone surface to volume ratio (BS/TV), calculated from the microCT reconstructions of the bone core biopsy samples. | 3-6 months
  Ratio of the segmented bone surface to the total volume in the region of interest. Unit: 1/mm
Value of the trabecular thickness (Tb.Th.), calculated from the microCT reconstructions of the bone core biopsy samples. | 3-6 months
  Mean thickness of the trabeculae, assessed using direct 3D methods. Unit: mm
Value of the trabecular separation (Tb.Sp.), calculated from the microCT reconstructions of the bone core biopsy samples. | 3-6 months
  Mean distance between the trabeculae, assessed using direct 3D methods. Unit: mm
Value of the trabecular bone pattern factor (Tb.Pf), calculated from the microCT reconstructions of the bone core biopsy samples. | 3-6 months
  Indicator of the relation between convex and concave elements in the trabecular bone structure. Tb.Pf <0 when the trabecular bone is honeycomb-like and increases as the trabecular bone acquires a rod-like structure. Unit: none
Value of the structure model index (SMI), calculated from the microCT reconstructions of the bone core biopsy samples. | 3-6 months
  The estimator of the plate- versus rod-like characteristic of the trabecular bone structure, 0 for perfect plates, 3 for perfect rods, and 4 for perfect spheres. Unit: none
Value of the Total porosity (Po(tot)), calculated from the microCT reconstructions of the bone core biopsy samples. | 3-6 months
  Percent porosity is the volume of pores as a percent of the total volume of interest (VOI). Unit: percent (%)
Value of the Connectivity (Conn.), calculated from the microCT reconstructions of the bone core biopsy samples. | 3-6 months
  One useful and fast algorithm for calculating the Euler connectivity in 3D is the "Conneulor". It measures what might be called "redundant connectivity", the degree to which parts of the object are multiply connected. It is a measure of how many connections in a structure can be severed before the structure falls into two separate pieces. Unit: none.

CONTACTS AND LOCATIONS:
Overall Officials: Márton Kivovics, DMD,MSD,PHD, Principal Investigator — Department of Public Dental Health, Semmelweis University
Locations (1):
- Semmelweis University Department of Public Dental Health, Budapest, Budapest, Hungary

IPD SHARING:
Plan to Share IPD: No